CLINICAL TRIAL: NCT02024399
Title: Pilot Study of 10 Week Exercise and Nutrition Program for Children Who Are Overweight / Obese.
Brief Title: Cardiovascular Risk Factors, Body Composition, Fitness Levels And Quality Of Life In Overweight And Obese 8-17 Year Olds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 87468
Record Dates: First submitted 2013-12-26; First posted 2013-12-31 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Childhood Obesity; Type 2 Diabetes; Hypercholesterolemia; Hypertension
Keywords: Pediatric Overweight/Obesity, DEXA, Fitness
MeSH Terms: conditions — Pediatric Obesity; Diabetes Mellitus, Type 2; Hypercholesterolemia; Hypertension; Obesity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exercise (Other): Strength training x 20 sessions (10 weeks) Aerobic exercise core strengthening Running
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Strength training, aerobic exercise and core strengthening, running

SUMMARY:
This project will address the important area of childhood obesity and the risk of cardiovascular disease associated with obesity. This is a serious health concern since children who are overweight or obese are prone to other medical conditions including high blood pressure, abnormal lipid profiles,and type 2 diabetes. Although exercise and nutrition programs are recommended, evidence for the efficacy of these programs in improving cardiovascular health is lacking.

Specific Aims: a) improve cardiovascular risk factors, b) increase physical fitness levels, c) improve lean body mass, d) enhance QOL of the child e) influence adherence rates to exercise and a healthy lifestyle change both during and beyond the conclusion of the program.

Hypothesis 1a: Compared to baseline and matched controls, children randomized to a 10 week multidisciplinary fitness and nutrition program will show significant improved levels of cardiovascular risk factors.

Specific Aim 2: To determine if a multidisciplinary fitness and nutrition program, when compared with a matched, WLC group will show a change in whole body assessment including a decrease in fat mass, an increase in percent lean body mass, and a decrease in percent body fat, as measured utilizing dual-energy X-ray absorptiometry Hypothesis 2a: Compared to baseline and matched controls, children randomized to a 10 week multidisciplinary fitness and nutrition program will show improved whole body assessments including.

Specific Aim 3:To determine if a multidisciplinary fitness and nutrition program, when compared with a WLC group will show improved levels of fitness. Hypothesis 3a: Compared to baseline and matched controls, children randomized to a 10 week multidisciplinary fitness and nutrition program will show significant improvements in fitness including.

ELIGIBILITY:
Inclusion Criteria:

* : a) in the 85th percentile Body Mass Index(BMI), standardized for age and gender; b) have hypercholesterolemia as defined as total cholesterol > 170 mg/dl or LDL > 110 mg/dl; and / or c) hypertension as defined as >116/76 for 8-10 year olds, > 120/80 for 10-13 year olds, and >125/890 for 14-17 year olds.

Exclusion Criteria:

* 1) age < 8 or > 17 years; 2) the determination of significant abnormalities on an initial graded exercise test performed by a pediatric cardiologist; 3) past history of chemotherapy or whole-body radiation therapy

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2004-08; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Improved body compositon (decrease in % fat; increase in % lean tissue) using DEXA | Baseline, after 10 weeks and after 20 weeks (3 time points)
  Dual energy x-ray absorptiometry - used to assess body composition.

SECONDARY OUTCOMES:
Improved levels of fitness using ACSM guidelines / assessments to measure such constructs of fitness as flexibility, muscle strength, cardiovascular endurance and agility. | Measured at baseline, after 10 week sand again after 20 weeks.
  ACSM guidelines and measurement were used to assess strength, agility, flexibility, muscle endurance and cardiovascular endurance

OTHER OUTCOMES:
Quality of life as perceived by the children and the parents. | Baseline and after 10 weeks and 20 weeks.
  The impact of weight on quality of life was utilized.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon A Martino, PhD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University, Stony Brook, New York, United States